CLINICAL TRIAL: NCT00008736
Title: Electrogastrography (EGC) in Premature Infants With Feeding Intolerance: The Effect of Metoclopramide
Brief Title: Electrogastrography (EGC) in Premature Infants With Feeding Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR00240-1724
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Infant, Newborn, Diseases
Keywords: Feeding intolerance; Infant, premature
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth | interventions — Metoclopramide

INTERVENTIONS:
Drug: metoclopramide

SUMMARY:
Serial EGC measurements in premature infants attempting to correlate EGC measurements with signs of feeding intolerance and response to metoclopramide therapy.

ELIGIBILITY:
Inclusion:

Premature infants. Absence of 1) infection, 2) congenital anomalies, 3) growth retardation

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States